CLINICAL TRIAL: NCT02223741
Title: An Observational Study of the Conventional Rehabilitation and Traditional Korean Medicine Conjugated Rehabilitation on Children With Cerebral Palsy
Brief Title: Observational Study of the Conjugated Rehabilitation on Children With Cerebral Palsy
Status: Completed | Type: Observational
Sponsor: Korean Medicine Hospital of Pusan National University (Other)
Collaborators: Korea Health Industry Development Institute (Other Government)
Responsible Party: Principal Investigator, Young Ju Yun, Associate Professor, Korean Medicine Hospital of Pusan National University
Other Study IDs: CP_conjugated rehabilitation
Record Dates: First submitted 2014-08-20; First posted 2014-08-22 (Estimated); Last update posted 2020-02-25 (Actual); Status verified 2020-02

CONDITIONS: Cerebral Palsy
Keywords: Cerebral palsy; GMFM-66; PEDI
MeSH Terms: conditions — Cerebral Palsy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 12 Months
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Korean medicine conjugate rehabilitation: those with more than 30 days of herbal drugs or more than 12 times of acupuncture (Korean medical treatment) within six months in addition to conventional rehabilitation
  Interventions: Other: Korean medical treatment
- Conventional rehabilitation: those with one of the treatments; physical, occupational, speech-language or cognitive-behavioral therapies

INTERVENTIONS:
Other: Korean medical treatment — acupuncture and herbal drugs
  Groups: Korean medicine conjugate rehabilitation

SUMMARY:
This study is designed to assess effectiveness, safety and cost-utility of conventional rehabilitation and traditional Korean medicine conjugated rehabilitation on children with cerebral palsy.

DETAILED DESCRIPTION:
1. Survey

   1. An interview survey on baseline

      * Basic characteristics
      * Cause of cerebral palsy
      * Accompanied disorders
      * Health problems
      * Operation history
      * Drug-taking
      * Rehabilitation treatment
      * Korean medicine treatment
      * Health functional food
      * Medical care cost
   2. An interview survey on 26th and 52nd weeks

      * Accompanied disorders
      * Health problems
   3. A weekly tracking survey

      * Health problems
      * Therapeutic change
      * Medical care cost
      * Quality of life
2. Assessment for function development on baseline, 26th and 52nd weeks

   * Gross Motor Function Classification System (GMFCS)
   * Gross Motor Function Measure-66 (GMFM-66)
   * Pediatric Evaluation of Disability Inventory (PEDI)

ELIGIBILITY:
Inclusion Criteria:

* Children with cerebral palsy
* Age from 6 to 78 months
* whose guardian consent to the present study

Exclusion Criteria:

* who had an orthopedic operation due to cerebral palsy
* who has congenital muscular disease, hereditary disease, or progressive central nervous system diseases
* who suffers from severe diseases (ie, cancer, severe heart disease, severe infectious disease)

Ages: 6 Months to 78 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Population will be selected from rehabilitation clinics for children
Sampling Method: Non-Probability Sample
Enrollment: 207 (Actual)
Dates: Start 2014-08 (Actual); Primary Completion 2017-05-11 (Actual); Study Completion 2017-05-11 (Actual)

PRIMARY OUTCOMES:
Change from baseline on GMFM-66 scores at week 26 and 52 | Baseline, Week 26, Week 52
  The GMFM-66 includes 66 items identified through Rasch analysis, which, together, best describe gross motor function in children with cerebral palsy of varying abilities.
Change from baseline on PEDI scores at week 26 and 52 | Baseline, Week 26, Week 52
  The PEDI measures abilities in the three functional domains of self-care, mobility and social function with 217 questions.

SECONDARY OUTCOMES:
Change of severity from baseline on accompanied disorders and health problems at week 24 and 52 | Baseline, Week 26, Week 52

OTHER OUTCOMES:
Economy evaluation | Baseline, Week 26, Week 52
  Direct and indirect medical care cost, Labor productivity of family
Number of Participants with Serious and Non-Serious Adverse Events | up to 52 weeks
Change from baseline on height and weight at week 24 and 52 | Baseline, Week 26, Week 52

CONTACTS AND LOCATIONS:
Overall Officials: Young-Ju Yun, MD, Ph D., Principal Investigator — Pusan National University Korean Medicine Hospital
Locations (6):
- South Korea (6):
  - Pusan national University Yangsan Hospital, Yangsan, Gyeongsangnam-do
  - Pusan National University Hospital, Busan
  - Seongmo-i Oriental Medical Clinic, Daegu
  - Haema Oriental Medical Clinic, Seoul
  - Heoyoungjin Oriental Medical Clinic, Seoul
  - Dong-Eui University Korean Medical Hospital, Ulsan

REFERENCES:
- [Derived] Yoo JE, Yun YJ, Shin YB, Kim NK, Kim SY, Shin MJ, Yu SA. Protocol for a prospective observational study of conventional treatment and traditional Korean medicine combination treatment for children with cerebral palsy. BMC Complement Altern Med. 2016 Jun 8;16:172. doi: 10.1186/s12906-016-1161-6. PMID 27267182